CLINICAL TRIAL: NCT05653999
Title: Assessing Speech Perception and Amplification Benefit During Infancy
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Sonova AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 22-2169
Record Dates: First submitted 2022-12-02; First posted 2022-12-16 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss; Children With Hearing Differences; Amplification; Speech Perception
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Normal Hearing: Group 1 will consist of approximately 20 infants with normal hearing. This cohort will have passed their newborn hearing screenings and will pass audiologic measurements on the day of testing. Audiologic measurements include tympanometry to determine middle ear function and otoacoustic emissions testing to determine cochlear integrity.
- Hearing Loss: Group 2 will consist of approximately 20 infants with diagnosed bilateral sensorineural hearing loss ranging from mild to severe. These infants will also pass audiologic measures on the day of testing (tympanometry as described in group 1), currently use bilateral air-conduction hearing aids, and are enrolled in early intervention services.
  Interventions: Device: Hearing Aids

INTERVENTIONS:
Device: Hearing Aids — Hearing aids will be used by infants with a diagnosed sensorineural hearing loss.
  Groups: Hearing Loss

SUMMARY:
The goal of this project is to compare aided and unaided speech discrimination among infants with hearing loss and a cohort of infants with typical hearing.

Working Hypothesis: Among this group of infants with hearing loss, performance will be significantly better when infants are tested while using amplification (i.e., aided condition) compared to when tested without amplification (i.e., unaided condition). Infants fit with optimally programmed amplification will perform similarly to the infants with typical hearing on speech discrimination tasks.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 months and 36 months (inclusive) at the time of enrollment.
* English is the primary spoken language in the home
* Demonstrated ability to complete a conditioned head turn via visual reinforcement audiometry (VRA)
* If normal hearing

  -Normal hearing sensitivity bilaterally
* If Hearing Loss

  * Children with diagnosis of bilateral sensorineural hearing ranging from mild to severe
  * Children currently using hearing aids
  * Children currently enrolled in intervention

Exclusion Criteria:

* Children born earlier than 35 weeks gestation
* Children with abnormal tympanometry on the day of testing
* Children with concerns of secondary disabilities
* Children with Auditory Neuropathy
* Concerns of hearing loss in normal hearing children

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants between 6 and 36 months of age (inclusively) will be be enrolled in either the normal hearing or hearing loss cohort based on hearing status. Infants will be recruited from the community as well as through established clinical relationships with the principal investigator at Children's Hospital Colorado Audiology Centers.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Behavioral Speech Perception | Through study completion, up to 6 weeks pending subject factors (e.g., fatigue, otitis media)
  To measure speech perception ability, infants are trained to complete a task in response to a change in a speech sound played over a speaker. Scores are given in d' (or equivalent) and are calculated from both true and false responses. Scores can range from 0.97 and 3.00. Scores above 1.2 are considered significantly above chance indicating successful perception of speech contrasts. To separate issues such as speech discrimination abilities versus proper conditioning, if a child is unable to discriminate a speech contrast (e.g., /ba-da/ or /sa-sha/) testing will transition to the 'easier' speech contrast /a-i/. If the child can discriminate between /a-i/, the investigators will repeat the previously tested contrast. Upon completion of this contrast the next contrast in will be assessed based on randomization ordering. If either contrast was not assessed/the child did not reach criterion, the participant will be rescheduled within 1 month, pending subject factors.

SECONDARY OUTCOMES:
Aided Behavioral Speech Perception Improvement | Through study completion, up to 6 weeks pending subject factors (e.g., fatigue, otitis media)
  Scores are measured from 0 to 2.03. Higher scores indicate greater benefit from hearing aid use in the hearing loss cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin M Uhler, PhD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado School of Medicine - Speech Perception Over Time Lab, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will review requests for de-identified data and review with appropriate regulatory bodies.